CLINICAL TRIAL: NCT00302640
Title: Multi-center, Double-blind, Placebo-controlled Study of Nitazoxanide Suspension in the Treatment of Diarrhea Caused by Enteric Viruses in Children
Brief Title: Study of Nitazoxanide Suspension in the Treatment of Diarrhea Caused by Enteric Viruses in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RM02-3021
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Rotavirus Infection; Adenoviridae Infection; Norovirus Infection
MeSH Terms: conditions — Rotavirus Infections; Adenoviridae Infections; Caliciviridae Infections | interventions — nitazoxanide

ARMS (2):
- Nitazoxanide (Active Comparator): 7.5mg/kg (age under 12 months), 5 mL (100mg nitazoxanide; age 1-3 years), 10 mL (200mg nitazoxanide; age 4-11 years) twice daily x 3 days
  Interventions: Drug: Alinia (nitazoxanide)
- Placebo (Placebo Comparator): 7.5mg/kg (age under 12 months), 5 mL (100mg nitazoxanide; age 1-3 years), 10 mL (200mg nitazoxanide; age 4-11 years) twice daily x 3 days
  Interventions: Drug: Alinia (nitazoxanide)

INTERVENTIONS:
Drug: Alinia (nitazoxanide)

SUMMARY:
The purpose of this study is to determine the effect of nitazoxanide suspension in treating diarrhea caused by enteric viruses in children less than 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Age <12 years.
* Patients with diarrhea (defined as 3 or more stools per day with liquid or semi-solid consistency, the number and consistency of stools being unusual for that person).
* Stool positive for adenovirus, norovirus or rotavirus by ELISA.

Exclusion Criteria:

* Females who are pregnant, suspected of being pregnant or breastfeeding.
* Other identified causes of diarrhea at screening.
* Serious systemic disorders incompatible with the study.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2005-02; Study Completion 2005-09

PRIMARY OUTCOMES:
Time from first dose to resolution of symptoms. | P-0.0105
  Median time: 31 hours for nitazoxanide group and 75 hours for the placebo group

SECONDARY OUTCOMES:
Virologic response (negative ELISA) at day 7-10.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Abu-Zekry, MD, Principal Investigator — Cairo University Children's Hospital, Cairo, Egypt

REFERENCES:
- [Result] Rossignol JF, Abu-Zekry M, Hussein A, Santoro MG. Effect of nitazoxanide for treatment of severe rotavirus diarrhoea: randomised double-blind placebo-controlled trial. Lancet. 2006 Jul 8;368(9530):124-9. doi: 10.1016/S0140-6736(06)68852-1. PMID 16829296